CLINICAL TRIAL: NCT05159895
Title: A Phase 1, Single-Center, Nonrandomized, Open-label Pharmacokinetic and Mass Balance Study of Oral-Administrated [14C]-DZD9008 in Healthy Male Subjects
Brief Title: Pharmacokinetic and Mass Balance Study of Oral-Administrated [14C]-DZD9008 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dizal Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DZ2021E0003
Record Dates: First submitted 2021-11-22; First posted 2021-12-16 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [14C]-DZD9008 (Experimental): A Single dose of [14C]-DZD9008
  Interventions: Drug: [14C]-DZD9008

INTERVENTIONS:
Drug: [14C]-DZD9008 — Each subject will receive a total of 100 mg DZD9008 oral suspension containing approximately 1 μCi of [14C] as a single administration

SUMMARY:
This is a phase 1, open-label, ADME study with single oral administration of [14C]-DZD9008 in healthy subjects.

DETAILED DESCRIPTION:
Phase 1 study to evaluate the excretion of DZD9008 radioactive dose, the metabolic profile, pharmacokinetics, safety and tolerability following a single oral administration of [14C]-DZD9008 in healthy male subjects. The purpose of this study is to investigate ADME properties of DZD9008 by analyzing blood, urine and feces samples collected during the study

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects between 18 and 60 years of age, with body mass index of 18.0 to 30.0 kg/m2. Body weight: ≥55 kg,and ≤ 100 kg.
* In good health, determined by no clinically significant findings from medical history, physical examination, 12-lead ECG, vital sign measurements, clinical laboratory evaluations.
* Regular bowel movements (ie, average production of ≥ 1 or ≤ 3 bowel movements a day).
* Adhere to specific contraception requirements
* Creatinine clearance ≥ 90 mL/min/1.73 m2.
* Aspartate aminotransferase and alanine aminotransferase must be ≤2.5 × upper limit of normal (ULN) and total bilirubin ≤1.5 × ULN.

Exclusion Criteria:

* Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, GI, neurological, respiratory, endocrine, or psychiatric disorder.
* History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the investigator, or history of hypersensitivity to DZD9008, its excipients, or drugs with a similar chemical structure or class.
* History of stomach or intestinal surgery history or presence of hepatic or renal disease or surgical procedure that would potentially alter absorption and/or excretion of orally-administered drugs (uncomplicated appendectomy and hernia repair will be allowed; cholecystectomy will not be allowed).
* Any clinically significant abnormalities in physical examination performed at check-in, vital signs (supine systolic blood pressure >140 mmHg, diastolic blood pressure >90 mmHg, and pulse rate ≥100 or ≤35 beats per minute) or clinical laboratory evaluations as judged by the investigator (or designee).
* Any clinically important abnormalities in rhythm, conduction, or morphology of resting 12-lead ECG, QTcF interval >450 msec, as judged by the investigator (or designee).
* A history of additional risk factors for Torsades de pointes (eg, heart failure, hypokalemia, family history of Long QT syndrome).
* Positive/reactive results on screening tests for serum hepatitis B surface antigen, hepatitis C antibody, or human immunodeficiency virus (Appendix 2).
* Acute illness, surgical procedures or trauma from within 2 weeks before screening until the first administration of the IMP.
* Subjects with active malignancy or neoplastic disease in the previous 12 months.
* Ongoing or planned inpatient surgery, dental procedure, or hospitalization during the study.
* Administration of a coronavirus disease 2019 (COVID-19) vaccine in the past 30 days prior to dosing.
* Use or intend to use any medications/products known to alter drug AME processes, including St. John's wort, within 30 days prior to check-in, unless deemed acceptable by the investigator (or designee).
* Use or intend to use any prescription medications/products within 28 days prior to check-in, unless deemed acceptable by the investigator (or designee). Exceptions may be allowed on a case by case basis as agreed by the investigator and sponsor's medical monitor if considered not to interfere with the aims of the study.
* Use or intend to use slow-release medications/products considered to still be active within 14 days prior to check-in, unless deemed acceptable by the investigator (or designee).
* Use or intend to use any nonprescription medications/products including vitamins, minerals, and phytotherapeutic/herbal/plant-derived preparations, gastric pH modifiers, and neutralizing antacids within 7 days prior to check-in, unless deemed acceptable by the investigator (or designee).
* Subjects will avoid the use of any prescription or nonprescription medications/products or herbal remedies that are strong/moderate CYP3A inhibitors or inducers within 28 days prior to check-in through the end of study, unless deemed acceptable by the Investigator.
* Subjects will avoid the use of any prescription or nonprescription medications/products or herbal remedies that are transporter (eg, P-gp) inhibitors or inducers within 28 days prior to the check-in through the end of study, unless deemed acceptable by the Investigator.
* Subjects should avoid the use of proton pump inhibitors from 7 days prior to check-in through 5 days postdose. For H2-antagonists or antacids, administration will follow the staggered schedule per protocol.
* Subjects who received a live or live-attenuated vaccine in the 2 weeks prior to IMP administration.
* Participation in a clinical study involving administration of an investigational drug (new chemical entity defined as a compound which has not been approved for marketing) or participation in any other clinical study (including methodology studies where no drugs were given) in the past 90 days prior to dosing.
* Subjects who have participated in any radiolabeled drug studies in the last 12 months prior to check-in.
* Have previously completed or withdrawn from this study or any other study investigating DZD9008 and have previously received DZD9008.
* History of alcohol abuse or excessive alcohol consumption, defined as > 21 units per week for males. One unit of alcohol equals 8.5 oz (250 mL) beer, 0.85 oz (25 mL) liquor, or 2.4 oz (125 mL) wine.
* Positive urine drug detected at screening, positive urinary alcohol test result or positive urine drug detected at check-in.
* History or suspected history of alcoholism or drug/chemical abuse within 2 years prior to check-in, as judged by the investigator (or designee).
* Use of tobacco- or nicotine-containing products within 3 months prior to check-in, or positive cotinine at screening or check-in.
* Ingestion of poppy seed-, Seville orange-, or grapefruit-containing foods or beverages within 7 days prior to check-in.
* Receipt of blood products within 2 months prior to check-in.
* Donation of blood from 3 months prior to screening, plasma from 2 weeks prior to screening, platelets from 6 weeks prior to screening, or any blood loss greater than 500 mL during the 3 months prior to screening.
* Poor peripheral venous access.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2021-09-24 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Percentage of Total Radioactivity (Cum% Dose) Recovered in Urine Relative to the Administered Radioactive Dose | Up to 85 days
Percentage of Total Radioactivity (Cum% Dose) Recovered in Feces Relative to the Administered Radioactive Dose | Up to 85 days
Amount of Total Radioactivity Excreted in Urine (Ae [UR]) | Up to 85 days
Amount of Total Radioactivity Excreted in Feces (Ae [Fe]) | Up to 85 days
Percentage of Administered Radioactive Dose (%Dose) Excreted in Urine for [14C]-DZD9008 | Up to 85 days
Percentage of Administered Radioactive Dose (%Dose) Excreted in Feces for [14C]-DZD9008 | Up to 85 days

CONTACTS AND LOCATIONS:
Overall Officials: Blanchard, Principal Investigator — Covance
Locations (1):
- Labcorp Clinical Research Unit, Madison site, Madison, Wisconsin, United States